CLINICAL TRIAL: NCT04357756
Title: A First-in-human (FIH), Open-Label, Phase I Dose Escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics of YH001 in Combination With Toripalimab Injection in Subjects With Advanced Solid Tumors
Brief Title: A Study to Assess YH001 in Combination With Toripalimab Injection in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eucure (Beijing) Biopharma Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YH001002
Record Dates: First submitted 2020-04-17; First posted 2020-04-22 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Advanced Solid Tumor
Keywords: dose escalation; safety; tolerability; advanced solid tumors; pharmacokinetics
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YH001 combined with Toripalimab (Experimental): All the patients will receive YH001 intravenously as single agent for 21 days followed by combination phase.
  Interventions: Drug: YH001; Drug: Toripalimab

INTERVENTIONS:
Drug: YH001 — YH001 will be administered intravenously every three weeks (Q3W) for 15 weeks (5 cycles) at doses of Dose A, Dose B, Dose C, Dose D, Dose E, Dose F and Dose G.
Drug: Toripalimab — Toripalimab will be administered by intravenously (Q3W) by the fixed dose of 240 mg from the 2nd cycle to 5th cycle.

SUMMARY:
This is an open-label, dose-escalation study of YH001 administered intravenously (IV) in combination with Toripalimab. The study is designed to determine the safety, tolerability and maximum tolerated dose (MTD) or recommended Phase 2 dose (RP2D) of YH001 when administered in combination with Toripalimab to subjects with advanced solid tumors.

DETAILED DESCRIPTION:
This trial will have a run-in phase to explore the safety and tolerability of YH001 as a single agent for 21 days as DLT observation period then followed by a combination phase to further explore the safety and tolerability of YH001 combined with Toripalimab (anti-PD-1 antibody) for each dose level during dose escalation.

The dose escalation will follow the traditional "3 + 3" dose escalation scheme. These subjects will be treated with YH001 and Toripalimab. YH001 will be administered intravenously every three weeks (Q3W) for 15 weeks (5 cycles) at doses of Dose A, Dose B, Dose C, Dose D, Dose E, Dose F and Dose G. Toripalimab will be administered by IV (Q3W) by the fixed dose of 240 mg from the 2nd cycle to 5th cycle. A single subject will be enrolled at Dose A as starting dose of YH001, and subsequent cohort will be expanded to include 3-6 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged ≥ 18 years
* Have advanced histologically or cytologically confirmed solid tumor
* Have progressed on after treatment with standard therapies or intolerant of standard care
* At least 1 unidimensional measurable target lesion per RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status score 0 or 1
* Have life expectancy of at least 12 weeks based on investigator's judgement

Exclusion Criteria:

* Treated with any investigational drug within 4 weeks prior to the fist dose of study drug
* Received any anticancer therapy less than 28 days prior to the first administration of study drug or within 5 half-lives of the therapy agent, whichever is shorter. Prior palliative radiotherapy to bone metastases ≤ 2 weeks prior to the first dose of YH001 is acceptable
* Subjects with prior anti-CTLA-4 checkpoint inhibitors should be excluded
* Subjects with prior PD-1/L1 treatment intolerate to PD-1/L1 therapy should be excluded
* Subjects with a history of ≥ Grade 3 immune-related adverse events (AEs) resulted from previous immunotherapy or an AE of any grade that resulted in discontinuation of prior immunotherapy
* Subjects with a history of ≥ Grade 2 pneumonitis resulted from previous immunotherapy or with a SpO2 by pulse oximetry < 92% at the screening
* Subjects requiring systemic treatment with corticosteroids (>10 mg/day prednisone or equivalent) or other immunosuppressive medications within 21 days before the planned first dose of study drug or has need to be treated while on trial. Inhaled or topical steroids, and adrenal replacement steroid doses ≤ 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease. Ophthalmologic, nasal and intra-articular injections of steroids are allowed
* Subjects with concomitant active autoimmune disease, history of autoimmune disease requiring systemic treatment, or history of autoimmune disease within the two years prior to study entry. Exceptions are subjects with vitiligo, resolved childhood asthma/atopy, type I diabetes mellitus or hypothyroidism which can be managed by replacement therapy
* Primary central nervous system (CNS) malignancies or symptomatic CNS metastases. But subjects with asymptomatic CNS metastases might be eligible if they have no clinical evidence of progression since completion of CNS-directed therapy, minimum 4 weeks between completion of radiotherapy and the first dose of YH001 and are currently not receiving corticosteroids
* QTc > 450 ms at baseline; no concomitant medications that would prolong the QT interval; no family history of long QT syndrome
* Continuance of toxicities due to prior radiotherapy or chemotherapy agents that have not recovered to ≤ Grade 1 per CTCAE v5.0, except alopecia, < Grade 2 sensory neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-04-21 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2022-10-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events and serious adverse events | From screening up to 1 year
  The safety profile of YH001 will be assessed by monitoring the adverse events (AE) per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0
Maximum tolerated dose (MTD) | During Cycle 1 (each cycle is 21 days)
  MTD is defined as the highest dose level at which no more than 1 out of 6 subjects experiences a DLT during the first cycle
Dose-limiting toxicities (DLT) | During Cycle 1 (each cycle is 21 days)
  DLT is defined as a toxicity (adverse event at least possibly related to YH001) occurring during the DLT observation period (the initial 21 days) both in run-in phase of YH001 as single agent and in combination phase of YH001 in combination with Toripalimab

SECONDARY OUTCOMES:
Area under the serum concentration versus time curve within one dosing interval (AUCtau) | Up to 1 year
  To determine the PK profile of YH001 alone and in combination with Toripalimab
Steady state AUC | Up to 1 year
  To determine the PK profile of YH001 alone and in combination with Toripalimab
Maximum serum concentration (Cmax) | Up to 1 year
  To determine the PK profile of YH001 alone and in combination with Toripalimab
Trough concentration before the next dose is administered (Ctrough) | Up to 1 year
  To determine the PK profile of YH001 alone and in combination with Toripalimab
Time to reach maximum serum concentration (Tmax) | Up to 1 year
  To determine the PK profile of YH001 alone and in combination with Toripalimab
Clearance (CL) | Up to 1 year
  To determine the PK profile of YH001 alone and in combination with Toripalimab
Volume of distribution (Vd) | Up to 1 year
  To determine the PK profile of YH001 alone and in combination with Toripalimab
Terminal half-life (T1/2) | Up to 1 year
  To determine the PK profile of YH001 alone and in combination with Toripalimab
Dose proportionality | Up to 1 year
  To determine the PK profile of YH001 alone and in combination with Toripalimab
Incidence of anti-drug antibodies (ADAs) | Up to 1 year
  To assess the immunogenicity of YH001 in combination with Toripalimab
Incidence of neutralizing antibodies (NAbs) | Up to 1 year
  To assess the immunogenicity of YH001 in combination with Toripalimab
Objective response rate (ORR) | Up to 1 year
  To assess the preliminary antitumor activity of YH001 in combination with Toripalimab
Duration of response (DOR) | Up to 1 year
  To assess the preliminary antitumor activity of YH001 in combination with Toripalimab
Time to response (TTR) | Up to 1 year
  To assess the preliminary antitumor activity of YH001 in combination with Toripalimab
Progression free survival (PFS) | Up to 1 year
  To assess the preliminary antitumor activity of YH001 in combination with Toripalimab
Overall survival (OS) | Up to 1 year
  To assess the preliminary antitumor activity of YH001 in combination with Toripalimab
Disease control rate (DCR) | Up to 1 year
  To assess the preliminary antitumor activity of YH001 in combination with Toripalimab
Duration of disease control (DDC) | Up to 1 year
  To assess the preliminary antitumor activity of YH001 in combination with Toripalimab

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Blacktown Hospital, Blacktown Cancer and Haematology Centre, Blacktown, New South Wales
  - St George Private Hospital, Kogarah, New South Wales
  - Peninsula & South Eastern Haematology and Oncology Group, Frankston, Victoria